CLINICAL TRIAL: NCT04556461
Title: Effects of Tralokinumab Treatment of Atopic Dermatitis on Skin Barrier Function
Acronym: TraSki
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dr. Stephan Weidinger (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Stephan Weidinger, Vice Head, University Hospital Schleswig-Holstein
Organization: University Hospital Schleswig-Holstein (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TRA-WEI-0015-I
Record Dates: First submitted 2020-07-16; First posted 2020-09-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Atopic Dermatitis
Keywords: Skin Barrier; Atopic Dermatitis; Dermatology; Biologics
MeSH Terms: conditions — Dermatitis, Atopic | interventions — tralokinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tralokinumab (Experimental): Tralokinumab 600mg loading dose s.c., followed by 300mg every other week.
  Interventions: Drug: Tralokinumab

INTERVENTIONS:
Drug: Tralokinumab — 2 x 300 mg Tralokinumab s.c. loading dose followed by 8 x 300 mg every 2 weeks (Q2W)

SUMMARY:
Effects of tralokinumab treatment of atopic dermatitis on skin barrier function.

DETAILED DESCRIPTION:
A phase II, monocenter , open, investigator initiated clinical trial investigating the effects of Tralokinumab treatment of atopic dermatitis on skin barrier physiology and function.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
2. Age ≥ 18 years at time of study entry.
3. Diagnosis of chronic atopic dermatitis for at least 1 year prior to enrollment based on American Academy Criteria
4. Subjects who have a recent history (within 1 year before the screening visit) of inadequate response to treatment with topical medications. Inadequate response is defined as failure to achieve and maintain remission or a low disease activity state (comparable to IGA 0=clear to 2=mild) despite treatment with a daily regimen of TCS of medium to higher potency (±TCI as appropriate), applied for at least 28 days or for the maximum duration recommended by the product prescribing information (e.g. 14 days for super-potent TCS), whichever is shorter. Subjects with documented systemic treatment for AD in the past year are also considered as inadequate responders to topical treatments and are potentially eligible for treatment with Tralokinumab after appropriate washout.
5. Eczema Area and Severity Index (EASI) score ≥12 at screening (Week0 minus 7d) and baseline visit (Week0)
6. Investigator Global Assessment (IGA) ≥3 at screening and baseline visit
7. Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial.
8. Female participants who are not capable of bearing children or who use a method of contraception that is medically approved by the health authority of the respective country at screening

   This includes:
   * A woman who is not capable of bearing a child is defined as follows: post-menopausal (12 months natural (spontaneous) amenorrhea or 6 months spontaneous amenorrhea with serum-FSH-values (follicle-stimulating hormone) of >40 mIU/mL); 6 weeks after a bilateral ovariectomy with or without hysterectomy or sterilization by means of tubal ligation
   * A woman capable of bearing child is defined as follows: a woman who is physiologically capable of becoming pregnant, including women whose occupation, lifestyle or sexual orientation exclude sexual intercourse with a male partner and women whose partners have been sterilized by vasectomy or other measures.
   * Medically-approved methods of contraception can include the following: hormonal contraceptives or, intrauterine device and double barrier method. Acceptable preventive measures can include total abstinence at the discretion of the investigator, in cases where compliance is ensured because of the study participant's age, occupation, lifestyle or sexual orientation. Periodical abstinence (e.g. calendar, ovulation, symptothermal methods or abstinence until the 4th day after the ovulation) as well as coitus interruptus are not acceptable methods of contraception.
   * A reliable method of contraception (CTFG guideline) must be used for the entire duration of the study.
9. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Subject is unable to provide written informed consent or comply with the protocol
2. Concurrent enrolment in another clinical trial where the subject is receiving an IMP or participation in another clinical trial with investigational product during the last 30 days before inclusion or 7 half-lives of previously used trial medication, whichever is longer.
3. Previous enrollment in a Tralokinumab clinical trial.
4. Active dermatologic conditions that may confound the diagnosis of AD or would interfere with assessment of treatment, such as scabies, cutaneous lymphoma, or psoriasis.
5. Known active allergic or irritant contact dermatitis that is likely to interfere with the assessment of severity of AD.
6. Subject with mild atopic dermatitis (EASI<12 and IGA<3) or is not a candidate or is not eligible for Tralokinumab treatment, because of a known or suspected allergy or reaction to any component of the IMP formulation or other possible contraindications like trypanophobia
7. Having used immunosuppressive/immunomodulating therapy (Systemic immunosuppressive/immunomodulating drugs (e.g. methotrexate, cyclosporine, azathioprine, mycophenolate mofetil, Janus kinase inhibitors), systemic corticosteroid use (excludes topical, inhaled, or intranasal delivery, bleach baths) during any week within the 4 weeks or tanning beds or phototherapy (narrow band ultraviolet B [NBUVB], ultraviolet B [UVB], ultraviolet A1 [UVA1], psoralen + ultraviolet A [PUVA]), within 4 weeks before the baseline visit
8. Treatment of selected skin areas (non-lesional skin at volar forearm and extensor forearm, lesional skin) with topical corticosteroid or topical calcineurin inhibitor 1 week prior to baseline visit and throughout the study.
9. Treatment of skin areas of examination with emollients 24 hours prior to baseline visit and throughout the study.
10. Involvement in the planning and/or conduct of the study.
11. Dementia or significantly altered mental status that would prohibit the understanding or rendering of information, consent and compliance with the requirements of the protocol and patients who are legally institutionalized.
12. Pregnancy and breastfeeding are exclusion factors. The effects of Tralokinumab on the developing human fetus are unknown. Enrolled patients must agree to use adequate contraception prior to study entry, the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
13. Medication that is known to interfere with any of the agents applied in the trial.
14. Receipt of live attenuated vaccines 30 days prior to the date of baseline and during the trial including the safety follow-up period.

    a. Receipt of inactive/killed vaccinations (e.g. inactive influenza) is allowed, provided they are not administered within 5 days before/after any trial visit.
15. Receipt of any marketed biological therapy (i.e. immunoglobulin, anti-IgE) including dupilumab or investigational biologic agents:

    1. Any cell-depleting agents including but not limited to rituximab: within 6 months prior to baseline or until lymphocyte count returns to normal whichever is longer.
    2. Other biologics: within 3 months or 5 half-lives, whichever is longer prior to baseline.
16. Receipt of any investigational non-biologic agent within 5 half-lives prior to baseline.
17. Receipt of blood products within 4 weeks prior to screening.
18. Major surgery within 8 weeks prior to screening, or planned in-patient surgery or hospitalization during the trial period.
19. History of any active skin infection within 1 week prior to baseline.
20. History of a clinically significant infection within 4 weeks prior to baseline which, in the opinion of the investigator or sponsor, may compromise the safety of the subject in the trial, interfere with evaluation of the IMP, or reduce the subject's ability to participate in the trial. Clinically significant infections are defined as:

    1. A systemic infection.
    2. A serious skin infection requiring parenteral (intravenous or intramuscular) antibiotics, antiviral, or antifungal medication.
21. History of a helminthic parasitic infection within 6 months prior to the date informed consent is obtained that has not been treated with, or has failed to respond to, standard of care therapy.
22. History of anaphylaxis following any biological therapy.
23. History of immune complex disease.
24. History of cancer:

    1. Subjects who have had basal cell carcinoma, localized squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible provided that the subject is in remission and curative therapy was completed at least 12 months prior to the date informed consent was obtained.
    2. Subjects who have had other malignancies are eligible provided that the subject is in remission and curative therapy was completed at least 5 years prior to the date informed consent was obtained.
25. History of tuberculosis requiring treatment within the 12 months prior to screening. Evaluation will be according to local guidelines as per local standard of care.
26. History of any known primary immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test at screening, or the subject taking antiretroviral medications as determined by medical history and/or subject's verbal report.
27. History of chronic alcohol or drug abuse within 12 months prior to screening, or any condition associated with poor compliance as judged by the investigator.
28. Any disorder, including but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, immunological, psychiatric, or major physical impairment that is not stable, in the opinion of the investigator, and could:

    1. Affect the safety of the subject throughout the trial.
    2. Influence the findings of the trial or their interpretations.
    3. Impede the subject's ability to complete the entire duration of trial.
29. Any clinically significant abnormal findings in physical examination, vital signs, hematology or clinical chemistry during the screening period, which in the opinion of the investigator, may put the subject at risk because of his/her participation in the trial, or may influence the results of the trial, or the subject's ability to complete entire duration of the trial.
30. Positive hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (HBsAb), hepatitis B core antibody (HBcAb) or hepatitis C virus antibody (anti-HCV) serology at screening.
31. Pregnant, breastfeeding, or lactating women.
32. Employees of the trial site or any other individuals directly involved

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Skin barrier function | 16 weeks
  Primary Endpoint is the change in transepidermal water loss (TEWL) at one non-lesional and one lesional marker skin area at week 16 (day 112) compared to baseline (day 0).

SECONDARY OUTCOMES:
Effect of tralokinumab treatment on skin irritability | 16 weeks
  Change in skin irritability: Change in clinical score of sodium lauryl sulfate irritant reaction of non-lesional skin at week 16 compared to baseline (Erythema, Infiltration/Edema, Squamation, Oozing/Crusting will be evaluated on a 4-point scale with non-existent (0) to severe (3))
Effect of Tralokinumab treatment on epidermal differentiation. | 16 weeks
  Change of epidermal thickness of one lesional and one non-lesional marker skin area at week 16 compared to baseline (μm)
Effect of tralokinumab treatment on disease activity. | 16 weeks
  Mean percent change at week 16 from baseline in Eczema Area and Severity Index (EASI) (values from 0 to 72 possible, where an EASI >12 indicates a moderate to severe disesase)

OTHER OUTCOMES:
Effect of tralokinumab treatment on the skin transcriptome. | 16 weeks
  Percent mean change of expression fold change of marker skin transcripts between AL and AN at week 16 as compared to baseline .
Effect of tralokinumab treatment on the skin proteome. | 16 weeks
  Percent mean change of expression fold change of marker skin proteins between AL and AN at week 16 as compared to baseline .
Effect of tralokinumab treatment on the skin microbiome. | 16 weeks
  Percent change in Shannon and Bray-Curtis index from baseline to week 16

CONTACTS AND LOCATIONS:
Locations (1):
- UKSH, Campus Kiel, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eichenfield LF, Ahluwalia J, Waldman A, Borok J, Udkoff J, Boguniewicz M. Current guidelines for the evaluation and management of atopic dermatitis: A comparison of the Joint Task Force Practice Parameter and American Academy of Dermatology guidelines. J Allergy Clin Immunol. 2017 Apr;139(4S):S49-S57. doi: 10.1016/j.jaci.2017.01.009. PMID 28390477
- [Background] Weidinger S, Novak N. Atopic dermatitis. Lancet. 2016 Mar 12;387(10023):1109-1122. doi: 10.1016/S0140-6736(15)00149-X. Epub 2015 Sep 13. PMID 26377142
- [Background] Bieber T. Atopic dermatitis. Ann Dermatol. 2010 May;22(2):125-37. doi: 10.5021/ad.2010.22.2.125. Epub 2010 May 17. PMID 20548901
- [Background] Silverberg JI, Hanifin JM. Adult eczema prevalence and associations with asthma and other health and demographic factors: a US population-based study. J Allergy Clin Immunol. 2013 Nov;132(5):1132-8. doi: 10.1016/j.jaci.2013.08.031. Epub 2013 Oct 4. PMID 24094544
- [Background] Hanifin JM, Reed ML; Eczema Prevalence and Impact Working Group. A population-based survey of eczema prevalence in the United States. Dermatitis. 2007 Jun;18(2):82-91. doi: 10.2310/6620.2007.06034. PMID 17498413
- [Background] Kiebert G, Sorensen SV, Revicki D, Fagan SC, Doyle JJ, Cohen J, Fivenson D. Atopic dermatitis is associated with a decrement in health-related quality of life. Int J Dermatol. 2002 Mar;41(3):151-8. doi: 10.1046/j.1365-4362.2002.01436.x. PMID 12010340
- [Background] Tazawa T, Sugiura H, Sugiura Y, Uehara M. Relative importance of IL-4 and IL-13 in lesional skin of atopic dermatitis. Arch Dermatol Res. 2004 Apr;295(11):459-64. doi: 10.1007/s00403-004-0455-6. Epub 2004 Mar 10. PMID 15014952
- [Background] Omori-Miyake M, Yamashita M, Tsunemi Y, Kawashima M, Yagi J. In vitro assessment of IL-4- or IL-13-mediated changes in the structural components of keratinocytes in mice and humans. J Invest Dermatol. 2014 May;134(5):1342-1350. doi: 10.1038/jid.2013.503. Epub 2013 Nov 26. PMID 24280725
- [Background] Tsoi LC, Rodriguez E, Degenhardt F, Baurecht H, Wehkamp U, Volks N, Szymczak S, Swindell WR, Sarkar MK, Raja K, Shao S, Patrick M, Gao Y, Uppala R, Perez White BE, Getsios S, Harms PW, Maverakis E, Elder JT, Franke A, Gudjonsson JE, Weidinger S. Atopic Dermatitis Is an IL-13-Dominant Disease with Greater Molecular Heterogeneity Compared to Psoriasis. J Invest Dermatol. 2019 Jul;139(7):1480-1489. doi: 10.1016/j.jid.2018.12.018. Epub 2019 Jan 11. PMID 30641038
- [Background] Aleksza M, Lukacs A, Antal-Szalmas P, Hunyadi J, Szegedi A. Increased frequency of intracellular interleukin (IL)-13 and IL-10, but not IL-4, expressing CD4+ and CD8+ peripheral T cells of patients with atopic dermatitis. Br J Dermatol. 2002 Dec;147(6):1135-41. doi: 10.1046/j.1365-2133.2002.05013.x. PMID 12452862
- [Background] Purwar R, Werfel T, Wittmann M. IL-13-stimulated human keratinocytes preferentially attract CD4+CCR4+ T cells: possible role in atopic dermatitis. J Invest Dermatol. 2006 May;126(5):1043-51. doi: 10.1038/sj.jid.5700085. PMID 16484990
- [Background] Oh MH, Oh SY, Lu J, Lou H, Myers AC, Zhu Z, Zheng T. TRPA1-dependent pruritus in IL-13-induced chronic atopic dermatitis. J Immunol. 2013 Dec 1;191(11):5371-82. doi: 10.4049/jimmunol.1300300. Epub 2013 Oct 18. PMID 24140646
- [Background] Zheng T, Oh MH, Oh SY, Schroeder JT, Glick AB, Zhu Z. Transgenic expression of interleukin-13 in the skin induces a pruritic dermatitis and skin remodeling. J Invest Dermatol. 2009 Mar;129(3):742-51. doi: 10.1038/jid.2008.295. Epub 2008 Oct 2. PMID 18830273
- [Background] Blauvelt A, de Bruin-Weller M, Gooderham M, Cather JC, Weisman J, Pariser D, Simpson EL, Papp KA, Hong HC, Rubel D, Foley P, Prens E, Griffiths CEM, Etoh T, Pinto PH, Pujol RM, Szepietowski JC, Ettler K, Kemeny L, Zhu X, Akinlade B, Hultsch T, Mastey V, Gadkari A, Eckert L, Amin N, Graham NMH, Pirozzi G, Stahl N, Yancopoulos GD, Shumel B. Long-term management of moderate-to-severe atopic dermatitis with dupilumab and concomitant topical corticosteroids (LIBERTY AD CHRONOS): a 1-year, randomised, double-blinded, placebo-controlled, phase 3 trial. Lancet. 2017 Jun 10;389(10086):2287-2303. doi: 10.1016/S0140-6736(17)31191-1. Epub 2017 May 4. PMID 28478972
- [Background] Simpson EL, Bieber T, Guttman-Yassky E, Beck LA, Blauvelt A, Cork MJ, Silverberg JI, Deleuran M, Kataoka Y, Lacour JP, Kingo K, Worm M, Poulin Y, Wollenberg A, Soo Y, Graham NM, Pirozzi G, Akinlade B, Staudinger H, Mastey V, Eckert L, Gadkari A, Stahl N, Yancopoulos GD, Ardeleanu M; SOLO 1 and SOLO 2 Investigators. Two Phase 3 Trials of Dupilumab versus Placebo in Atopic Dermatitis. N Engl J Med. 2016 Dec 15;375(24):2335-2348. doi: 10.1056/NEJMoa1610020. Epub 2016 Sep 30. PMID 27690741
- [Background] Wollenberg A, Howell MD, Guttman-Yassky E, Silverberg JI, Kell C, Ranade K, Moate R, van der Merwe R. Treatment of atopic dermatitis with tralokinumab, an anti-IL-13 mAb. J Allergy Clin Immunol. 2019 Jan;143(1):135-141. doi: 10.1016/j.jaci.2018.05.029. Epub 2018 Jun 12. PMID 29906525
- [Background] May RD, Monk PD, Cohen ES, Manuel D, Dempsey F, Davis NH, Dodd AJ, Corkill DJ, Woods J, Joberty-Candotti C, Conroy LA, Koentgen F, Martin EC, Wilson R, Brennan N, Powell J, Anderson IK. Preclinical development of CAT-354, an IL-13 neutralizing antibody, for the treatment of severe uncontrolled asthma. Br J Pharmacol. 2012 May;166(1):177-93. doi: 10.1111/j.1476-5381.2011.01659.x. PMID 21895629
- [Background] Thom G, Minter R. Optimization of CAT-354, a therapeutic antibody directed against interleukin-13, using ribosome display. Methods Mol Biol. 2012;805:393-401. doi: 10.1007/978-1-61779-379-0_22. PMID 22094818
- [Background] Blanchard C, Mishra A, Saito-Akei H, Monk P, Anderson I, Rothenberg ME. Inhibition of human interleukin-13-induced respiratory and oesophageal inflammation by anti-human-interleukin-13 antibody (CAT-354). Clin Exp Allergy. 2005 Aug;35(8):1096-103. doi: 10.1111/j.1365-2222.2005.02299.x. PMID 16120093
- [Background] Guttman-Yassky E, Bissonnette R, Ungar B, Suarez-Farinas M, Ardeleanu M, Esaki H, Suprun M, Estrada Y, Xu H, Peng X, Silverberg JI, Menter A, Krueger JG, Zhang R, Chaudhry U, Swanson B, Graham NMH, Pirozzi G, Yancopoulos GD, D Hamilton JD. Dupilumab progressively improves systemic and cutaneous abnormalities in patients with atopic dermatitis. J Allergy Clin Immunol. 2019 Jan;143(1):155-172. doi: 10.1016/j.jaci.2018.08.022. Epub 2018 Sep 5. PMID 30194992
- [Background] Piper E, Brightling C, Niven R, Oh C, Faggioni R, Poon K, She D, Kell C, May RD, Geba GP, Molfino NA. A phase II placebo-controlled study of tralokinumab in moderate-to-severe asthma. Eur Respir J. 2013 Feb;41(2):330-8. doi: 10.1183/09031936.00223411. Epub 2012 Jun 27. PMID 22743678
- [Background] Dawson M, Wollenberg A, Silverberg JI, et al. A Phase 2b Dose-Ranging Efficacy and Safety Study of Tralokinumab in Adult Patients with Moderate to Severe Atopic Dermatitis. Ski J Cutan Med. 2018. doi:10.25251/skin.2.supp.28
- [Background] Kozich JJ, Westcott SL, Baxter NT, Highlander SK, Schloss PD. Development of a dual-index sequencing strategy and curation pipeline for analyzing amplicon sequence data on the MiSeq Illumina sequencing platform. Appl Environ Microbiol. 2013 Sep;79(17):5112-20. doi: 10.1128/AEM.01043-13. Epub 2013 Jun 21. PMID 23793624
- [Background] Dobin A, Davis CA, Schlesinger F, Drenkow J, Zaleski C, Jha S, Batut P, Chaisson M, Gingeras TR. STAR: ultrafast universal RNA-seq aligner. Bioinformatics. 2013 Jan 1;29(1):15-21. doi: 10.1093/bioinformatics/bts635. Epub 2012 Oct 25. PMID 23104886
- [Background] Robinson MD, Oshlack A. A scaling normalization method for differential expression analysis of RNA-seq data. Genome Biol. 2010;11(3):R25. doi: 10.1186/gb-2010-11-3-r25. Epub 2010 Mar 2. PMID 20196867
- [Background] Law CW, Chen Y, Shi W, Smyth GK. voom: Precision weights unlock linear model analysis tools for RNA-seq read counts. Genome Biol. 2014 Feb 3;15(2):R29. doi: 10.1186/gb-2014-15-2-r29. PMID 24485249
- [Background] Ritchie ME, Phipson B, Wu D, Hu Y, Law CW, Shi W, Smyth GK. limma powers differential expression analyses for RNA-sequencing and microarray studies. Nucleic Acids Res. 2015 Apr 20;43(7):e47. doi: 10.1093/nar/gkv007. Epub 2015 Jan 20. PMID 25605792
- [Background] Baurecht H, Ruhlemann MC, Rodriguez E, Thielking F, Harder I, Erkens AS, Stolzl D, Ellinghaus E, Hotze M, Lieb W, Wang S, Heinsen-Groth FA, Franke A, Weidinger S. Epidermal lipid composition, barrier integrity, and eczematous inflammation are associated with skin microbiome configuration. J Allergy Clin Immunol. 2018 May;141(5):1668-1676.e16. doi: 10.1016/j.jaci.2018.01.019. Epub 2018 Feb 5. PMID 29421277
- [Background] Holm EA, Wulf HC, Thomassen L, Jemec GB. Instrumental assessment of atopic eczema: validation of transepidermal water loss, stratum corneum hydration, erythema, scaling, and edema. J Am Acad Dermatol. 2006 Nov;55(5):772-80. doi: 10.1016/j.jaad.2006.03.036. Epub 2006 Jun 13. PMID 17052481
- [Derived] Tandon R, Harder I, Stolzl D, Hubenthal M, Sander N, Hartmann J, Suhrkamp I, Fonfara M, Gerdes S, Weidinger S. Tralokinumab Treatment of Atopic Dermatitis Induces a Progressive Transcriptomic Response. J Invest Dermatol. 2025 Jul;145(7):1643-1652.e13. doi: 10.1016/j.jid.2024.12.005. Epub 2024 Dec 27. PMID 39733934